CLINICAL TRIAL: NCT06630104
Title: MC230818 Understanding the Mechanisms of Clonal and Non-Clonal Cytopenia Following CAR-T Therapy
Brief Title: Understanding the Mechanisms of Clonal and Non-clonal Cytopenia Following CAR-T Therapy for Multiple Myeloma or CD19+ Lymphoproliferative Disorder (LPD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC230818; NCI-2024-07738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-005734 (Other: Mayo Clinic Institutional Review Board); MC230818 (Other: Mayo Clinic)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lymphoproliferative Disorder; Multiple Myeloma
MeSH Terms: conditions — Lymphoproliferative Disorders; Multiple Myeloma | interventions — Specimen Handling; Chromatin Immunoprecipitation Sequencing; Follow-Up Studies; Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (bone marrow aspiration, CFU) (Experimental): Patients undergo bone marrow aspiration and hair, buccal, saliva sample collection up to 14 days prior to LD therapy. Patients undergo CFU on day 90 post-CAR-T therapy. Patients with unexplained cytopenia also undergo bone marrow aspiration for sequencing analysis on day 90 and at development of MN-pCT during CFU. Patients also undergo bone marrow aspiration at determination of clonal evolution or myeloid neoplasm if not done during on day 90.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Other: Electronic Health Record Review; Procedure: Follow-Up; Other: Genetic Counseling; Other: Genetic Testing

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo hair, buccal, and saliva sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Other: Electronic Health Record Review — Ancillary studies
Procedure: Follow-Up — Undergo CFU
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
Other: Genetic Counseling — Receive genetic counselor consultation
Other: Genetic Testing — Undergo sequencing analysis
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test

SUMMARY:
This clinical trial evaluates the impact of preexisting and therapy-emergent germline and somatic variants on cytopenia in patients with multiple myeloma or CD19 positive lymphoproliferative disorder (LPD) following chimeric antigen receptor T-cell (CAR-T) therapy. The most common adverse event after CAR-T therapy is lower than normal blood cells (cytopenia) and up to one third of patients experience cytopenia that last longer than 30 days post-infusion. Germline and somatic variants are changes in genes found using cancer genomic tests. Cancer genetic/genomic testing is a series of tests that find specific changes in cancer cells or in blood deoxyribonucleic acid. Identifying gene mutations may help identify the risk of cytopenia in patients with multiple myeloma or CD19 positive LPD following CAR-T therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the preexisting and therapy-emergent germline and somatic variants associated with an increased risk of clonal and non-clonal cytopenia following CAR-T cell therapy on research basis.

SECONDARY OBJECTIVE:

I. Characterize the baseline transcriptomic signature associated with non-clonal and clonal cytopenia following CAR-T therapy on research basis.

OUTLINE:

Patients undergo bone marrow aspiration and hair, buccal, and saliva sample collection up to 14 days prior to lymphodepleting (LD) therapy. Patients undergo clinical follow-up (CFU) on day 90 post-CAR-T therapy. Patients with unexplained cytopenia also undergo bone marrow aspiration for sequencing analysis on day 90 and at development of myeloid neoplasm post-cytotoxic therapies (MN-pCT) during CFU. Patients also undergo bone marrow aspiration at determination of clonal evolution or myeloid neoplasm if not done during on day 90.

Patients with unexplained cytopenia at day 90 are followed up every 90 days for up to 2 years until resolution. Patients without unexplained cytopenia are followed clinically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed diagnosis of multiple myeloma (MM) as defined in International Myeloma Working Group (IMWG) criteria or a CD19+ lymphoproliferative disorder (LPD) as defined by 2016 World Health Organization (WHO) classification
* Provide written informed consent
* Willingness to provide mandatory bone marrow aspirate specimens for correlative research. All bone marrow aspirate samples are collected during a clinical procedure
* Willingness to provide mandatory hair follicle specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide saliva and buccal samples for research

Exclusion Criteria:

* Ineligible for CAR-T therapy
* Patients diagnosed with myeloid neoplasm before CAR-T therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Pathogenic and likely pathogenic germline and somatic variants associated with increased risk | At baseline
  The count and percentage of patients with the presence of somatic or germline variants will be reported. The number, type, and function of somatic variants will also be reported.
Unexplained cytopenia | At day 90
  Unexplained cytopenia will be defined per World Health Organization (WHO)-5 as a combination of any of the following: hemoglobin < 12 g/dL in females, hemoglobin < 13 g/dL in males, absolute neutrophil count < 1.8 x 10^9/L and platelets < 150 x 10^9/L. Logistic regression will be used to identify the presence or absence of baseline germline and somatic mutations associated with unexplained cytopenia. An odds ratio and 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Development of myeloid neoplasm post-cytotoxic therapies (MN-pCT) | Up to 2 years
  Assessed as development of MN-pCT at any time following CAR-T infusion. MN-pCT is defined per The World Health Organization- Five Well-Being Index (WHO-5). The count and percentage of patients with the presence of somatic or germline variants will be reported. The number, type, and function of somatic variants will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mithun V. Shah, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials